CLINICAL TRIAL: NCT05737056
Title: Rheumatoid Purpura in Children: a Multicenter Observational Study of Pediatric Emergency Department Management and Follow-up by Primary Care Physicians
Acronym: PREEMS
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Other Study IDs: GHRMSA 1278; 2022-A02687-36 (Other: ANSM)
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Purpura
MeSH Terms: conditions — IgA Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children diagnosed with rheumatoid purpura at the pediatric emergency department: Children diagnosed with rheumatoid purpura from admission to the pediatric emergency department up to two years of follow-up by general practitioners after hospital discharge.
  Interventions: Other: Management of rheumatoid purpura

INTERVENTIONS:
Other: Management of rheumatoid purpura — Collection of data on the management in pediatric emergency departments (method of diagnosis, complementary examinations, proposed treatment, number of hospitalizations, follow-up after hospital discharge).

SUMMARY:
The main objective of this study is to describe the management of children with rheumatoid purpura from admission to the pediatric emergency room to follow-up by primary care physicians after hospital discharge.

DETAILED DESCRIPTION:
Secondary objectives The secondary objective is to assess general practitioners current knowledge and practice of the condition and potential barriers to monitoring and follow-up by general practitioners.

Conduct of research Children diagnosed with rheumatoid purpura within the past 2 years at the 3 participating sites will be included in the study if parental authority holders do not object.

Patients will be identified through the Medical Information Department of each hospital.

Parents will be contacted - first by mail, then by phone - to request permission to collect the child's medical data from medical records, and to retrieve information on the surveillance and follow-up of the disease by general practitioners up to two years after diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Underaged patient diagnosed with rheumatoid purpura during a visit to the pediatric emergencies of Mulhouse, Colmar and Strasbourg
* No objection to the study from the two holders of parental authority

Exclusion Criteria:

- Patient followed in the context of a genetic or malformative pathology, an immune deficiency, or a cancer

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be identified by the Medical Information Department of each site. The study will be conducted on patients who have been managed for rheumatoid purpura within the last two years at one of the three participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Compliance with the recommendations for the management of rheumatoid purpura | Up to two years after hospital discharge

SECONDARY OUTCOMES:
Knowledge assessment questionnaire regarding rheumatoid purpura | At the beginning of the study
  Evaluation of the knowledge and current practices of general practitioners regarding rheumatoid purpura and identification of the possible obstacles to management and follow-up in primary care, using an online survey

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpitaux Civils de Colmar, Colmar
  - Hôpital de Hautepierre, Strasbourg

REFERENCES:
- See also: Study results — https://ecrin.app.unistra.fr/search/notice/view/ecrin-ori-356390